CLINICAL TRIAL: NCT05821075
Title: Comparative Study Between Prednisolone, Cerebrolysin in the Treatment of Bell's Palsy
Brief Title: Efficacy of Prednisolone Versus Cerebrolysin in the Treatment of Bell's Palsy
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: October 6 University (Other)
Responsible Party: Principal Investigator, engy wahsh, LECTURER OF CLINICAL PHARMACY, October 6 University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRC-Ph-2211038
Record Dates: First submitted 2023-04-07; First posted 2023-04-20 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Bell Palsy
MeSH Terms: conditions — Bell Palsy | interventions — Prednisolone; cerebrolysin

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Prednisolone (Active Comparator)
  Interventions: Drug: Prednisolone
- Cerebrolysin (Active Comparator)
  Interventions: Drug: Cerebrolysin
- Prednisolone and Cerebrolysin (Active Comparator)
  Interventions: Drug: Prednisolone; Drug: Cerebrolysin

INTERVENTIONS:
Drug: Prednisolone — prednisolone 60mg tablet once daily for 5 days then tapering dose
  Arms: Prednisolone; Prednisolone and Cerebrolysin
Drug: Cerebrolysin — intramuscular Cerebrolysin 10 mg daily for 3 weeks
  Arms: Cerebrolysin; Prednisolone and Cerebrolysin

SUMMARY:
Bell's palsy, a peripheral facial nerve paresis, is the most common disorder of the facial nerve and one of the most common mononeuropathies.

Many patients with Bell's palsy will develop some complications such as synkinesis, crocodile tears and 'sweating' of the ear while eating Commonly used medications to treat Bell's palsy is Corticosteroids Cerebrolysin stimulates the regeneration of the nervous tissue with protective action we aim to study the efficacy of cerebrolycin in Bell's palsy

ELIGIBILITY:
Inclusion Criteria:

* unilateral acute facial palsy of no identifiable cause

Exclusion Criteria:

* Recurrent facial Bell's palsy
* Pregnancy
* Diabetes
* Epilepsy
* Severe hypertension,
* Renal or hepatic disease,
* Gastric or duodenal ulcer
* presence of acute otitis media or ipsilateral chronic otitis
* Recent head injury,
* psychiatric disease
* If there is any contraindications for corticosteroids

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-08-24 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
change in scores of the house Brackman grading system HB | at baseline, after 1 week, after 3 week
changes in scores of the Sunnybrook grading system. | at baseline, after 1 week, after 3 week

CONTACTS AND LOCATIONS:
Locations (1):
- October 6 university hospital, Giza, Egypt